CLINICAL TRIAL: NCT04045184
Title: Improving the Quality of Food Assistance for People Living With HIV and Diabetes
Brief Title: Food Assistance, Diabetes, and HIV
Acronym: BFED
Status: Withdrawn | Type: Observational
Why Stopped: Stored specimens unavailable due to being depleted for COVID-19 research. Study converted to retrospective observational study of clinic patients diabetes trends using EMR data.
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Amanda Willig, Primary Investigator, University of Alabama at Birmingham
Other Study IDs: IRB-300001424; P30DK079626 (NIH)
Record Dates: First submitted 2019-04-01; First posted 2019-08-05 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Diabetes; HIV/AIDS; FOOD SECURITY
MeSH Terms: conditions — Diabetes Mellitus; Acquired Immunodeficiency Syndrome | interventions — Food Assistance

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Stored serum will be analyzed for markers of glycemic control: glucose, insulin, glycosylated hemoglobin, and fructosamine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- B-FED: Clients of the Birmingham AIDS Outreach Food and Education Delivery (B-FED) program who are also patients at the 1917 Clinic.
  Interventions: Other: Food assistance
- non B-FED: Patients at the 1917 Clinic who have chosen not to participate in B-FED at this time.

INTERVENTIONS:
Other: Food assistance — This is an observational study of an existing community program. No intervention is provided beyond food assistance in the community program.
  Other Names: no food assistance
  Groups: B-FED

SUMMARY:
Diabetes prevalence is increasing among people living with HIV (PLWH), yet blood glucose control is less successful in this population who are also often food insecure. Food assistance programs often provide nutrient-poor foods. This proposal asses the feasibility of monitoring diabetes-related health outcomes among food insecure PLWH who are receiving food boxes higher in dietary protein and fiber and lower in simple carbohydrates.

DETAILED DESCRIPTION:
The objective of this investigation is to develop and assess a study protocol to evaluate the impact of food assistance on diabetes-related health outcomes in food insecure people living with HIV (PLWH). Compared to the general population, PLWH have increased risk for type 2 diabetes and worse glycemic control when using similar pharmaceutical treatments. Interventions to improve diet quality could thus have a clinically meaningful impact on diabetes treatment in this population. However, many PLWH are food insecure and rely on food assistance to meet basic nutrition needs. This proposal will determine the feasibility of a protocol to evaluate diabetes-related health outcomes in food insecure PLWH and diabetes who receive high protein, high dietary fiber food boxes from Birmingham AIDS Outreach. The study will consist of retrospective analysis of electronic medical record data and stored specimens, and prospective cross-sectional analysis of food security and diet quality in PLWH who do versus those who do not receive the food boxes.

Specific Aim 1: To determine the feasibility of recruiting, enrolling, and collecting dietary intake data from people living with HIV who are food insecure.

Specific Aim 2: To compare changes over twelve months in glycemic control, food security, and diet quality in B-FED participants compared to non-participating 1917 clinic patients.

This proposal aligns with the UAB Diabetes Research Center's goal to facilitate development of new methods to treat diabetes and its complications. The investigators will determine the effect size for scale-up of larger, longer-term assessment through an NIDDK-R18 grant to evaluate the real-world impact of B-FED on glycemic control and food security.

ELIGIBILITY:
Inclusion Criteria:

* CNICS participants aged 18 and over
* Currently prescribed antiretroviral therapy
* Have a diagnosis of diabetes, or documented hemoglobin A1c >7.0%, or glucose >125gm/dL

Exclusion Criteria:

* Not diagnosed with HIV
* PLWH who are not patients at 1917 Clinic
* Under age 18
* Pregnant women
* Recent cancer diagnosis Current serious illness or trauma Persons with an active secondary infection including tuberculosis or untreated Hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be patients at the UAB 1917 Clinic who are diagnosed with HIV and type 2 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-10-20 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of recruiting, enrolling from people living with HIV who are food insecure. | 1 year
  We will track the ability to recruit and enroll eligible participants in the study.
Change in diabetes-related health outcomes as measured by hemoglobin A1c. | 1 year
  Six months after program enrollment, B-FED participants will have improved glycemic control (lower hemoglobin A1c). Value will be measured using stored blood samples.
Compare food security among groups using the Food Security Questionnaire. | 1 year
  B-FED participants will report a higher prevalence of food security compared to clinic patients who do not participate in the program. This will be assessed at 1 time point using the validated 2-item Food Security Questionnaire to classify participants as food secure, low food security, or very low food security.

CONTACTS AND LOCATIONS:
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
IPD will only be available to the study PI and research coordinator. Only deidentified data will be shared with other investigators.

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT04045184/SAP_000.pdf